| 课题编号 | 患者姓名 | 患者姓名拼音字母 | 病例编号 | 知情 |
|------|------|----------|------|-----|
| | | | | 同意书 |

# 受试者知情同意书

敬爱的患者:

您将被邀请参加一项由福建医科大学附属第一医院神经内科王志强医生(0591-87982772)主持的关于**面肩肱型型肌营养不良症(Facioscapulohumeral Muscular Dystrophy,FSHD)**的观察性研究。此项目由科研课题资助进行。由于您是面肩肱型肌营养不良症患者/基因携带者或家系成员而被邀请加入此项研究。本知情同意书提供给您一些信息以帮助您决定是否参加此项临床研究。您参加本项研究是自愿的。本次研究已通过本研究机构伦理审查委员会审查,伦理委员会办公室电话0591-87981029。如果你同意加入此项研究,请您仔细阅读下列说明,如有疑问请向研究者提出。

## 研究目的:

面肩肱型肌营养不良症(Facioscapulohumeral Muscular Dystrophy,FSHD)是一类常染色体显性遗传神经肌肉变性疾病,分为 1 型(FSHD1)和 2 型(FSHD2)两种类型,主要表现为对称性或不对称性肌无力和肌萎缩,累及面肌、肩胛带肌和上臂肌群,向下进展累及躯干肌群和下肢肌群,部分患者出现不同程度的合并症。因该病存在高度家系间和家系内临床异质性,且表观遗传规律特殊,目前其基因型与临床表型的相关性并不明确,为评价其肌肉病变,了解其自然发展病程以研究其遗传规律,我们将建立面肩肱型肌营养不良症的队列登记研究,分析发病因素,为探究进一步治疗研究储备依据。

#### 研究过程和方法:

如果您同意参与这项研究,我们将对每位受试者进行编号,建立病历档案。研究过程中将由专业人员为您取样,例如抽取静脉血 10毫升,如有需要将进行肌肉活检诊断手术,收集手术过程中剩余的组织约 50毫克,并进行成纤维和成肌细胞的分离培养。您的样品仅用于面肩肱型肌营养不良症(FSHD)的队列登记研究。

## 研究可能的受益:

通过对您的临床症状、分子检测及肌肉 MRI 改变的研究,将推动对营养不良症的认识及治疗方式进展。

### 研究风险与不适:

您参与这项研究无需承担任何费用及压力,也不会给您造成额外的伤害。样本采集 将严格按照无菌要求操作,可能会有短暂的疼痛、局部青紫、晕针等反应。

#### 隐私问题:

如果您决定参加本项研究,您参加试验及在试验中的个人资料均属保密。您的血/皮肤/肌肉活检标本将以研究编号数字而非您的姓名加以标识。可以识别您身份的信息将不会透露给研究小组以外的成员,除非获得您的许可。所有的研究成员和研究申办方都被要求对您的身份保密。您的档案将保存在福建医科大学附属第一医院神经内科档案柜中,仅供研究人员查阅。为确保研究按照规定进行,必要时,政府管理部门或伦理审查委员会的成员按规定可以在研究单位查阅您的个人资料。这项研究结果发表时,也需要对保密方面进行承诺。

## 自由退出:

作为受试者,您可随时了解与本研究有关的信息资料和研究进展,自愿决定(继续)参加还是不(继续)参加。参加后您可以选择在任何时候要求退出研究,您的数据将不纳入研究结果,任何医疗待遇与权益不会因此而受到影响。如果继续参加研究会对您造成严重的伤害,研究者也将会中止研究的进行。但在参加研究期间,请您提供有关自身病史和当前身体状况以及参与其他研究的真实情况,若因没有遵守研究计划,或者发生与研究相关的损伤等其它原因,研究医师可以终止您继续参与本项研究。

## 知情同意签字:

我已经阅读了本知情同意书,并且我的医生已经将此次临床试验的目的、内容、风险和受益情况向我作了详细的解释说明,对我询问的所有问题也给予了解答,我对此项临床研究已经了解,我自愿参加本项研究,在无特殊情况下,尽可能完整的接受本次临床研究。

| 受试者签名: | 研究者签字: |
|---------------------|--------------------|
| 联系手机号: | 联系手机号: |
| 日期: 年 月 日 | 日期: 年 月 日 |
| (如果受试者无识字能力则需见证人签名, | 如果受试者无行为能力则需代理人同意) |
| 法定代理人/见证人签名: | _ 与受试者关系: |